CLINICAL TRIAL: NCT04418908
Title: Vascular Disease, Inflammation and Hormones in Women With Type 1 Diabetes
Brief Title: Estrogen, Diabetes, and Endothelial Function
Acronym: EDEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 10-0591
Record Dates: First submitted 2020-05-26; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — cetrorelix; LHRH, N-acetyl-(4-chlorophenylalanyl)(1)-(4-chlorophenylalanyl)(2)-tryptophyl(3)-arginyl(6)-alanine(10)-; Estradiol

STUDY DESIGN:
Intervention Model Description: Participants were randomized to either receiving a gonadotropin-releasing antagonist (GnRHant) with estradiol add-back (+E2) or placebo (+PL). Investigators and participants were blinded to randomization status until the study was completed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GnRHant + E2 (Active Comparator): Participants in this arm received GnRHant and a transdermal estradiol patch (0.075 mg/day) for a period of 1 week.
  Interventions: Drug: Cetrorelix acetate, 0.25 mg/day; Drug: Estradiol Patch, 0.025 Mg/24 Hours Weekly Transdermal Film, Extended Release
- GnRHant + PL (Placebo Comparator): Participants in this arm received GnRHant and a placebo patch for a period of 1 week.
  Interventions: Drug: Cetrorelix acetate, 0.25 mg/day; Drug: Placebo patch

INTERVENTIONS:
Drug: Cetrorelix acetate, 0.25 mg/day — All participants self-administered GnRHant daily between the baseline and follow-up visits (cetrorelix acetate, 0.25 mg/day).
  Other Names: Cetrotide; GnRHant
Drug: Estradiol Patch, 0.025 Mg/24 Hours Weekly Transdermal Film, Extended Release — Active estradiol transdermal patch.
  Other Names: Climara
  Arms: GnRHant + E2
Drug: Placebo patch — Placebo patch designed to match active Climara patches.
  Arms: GnRHant + PL

SUMMARY:
This study planned to learn more about women and how the drop in estradiol levels during menopause may affect their cardiovascular risk. With aging, the arteries that are located around the heart get stiffer, and this increase in arterial stiffness can lead to a number of health problems such as high blood pressure and heart disease. In this study, the investigators examined whether a short-term drop in estrogen levels caused arteries to become stiffer, and explored potential reasons for stiffening arteries.

DETAILED DESCRIPTION:
Participants completed two study visits. The baseline study visit occurred during the early follicular phase of the menstrual cycle, confirmed via take-home ovulation testing. On the day of the baseline study visit, all participants underwent ovarian sex hormone suppression with GnRHant therapy (cetrorelix acetate, 0.25 mg/day) delivered daily as subcutaneous injections for a 1-week period. Participants were randomized to one of two concurrent intervention groups: transdermal estradiol patch (0.075 mg/day) (+E2) or placebo patch (+PL) and returned for a follow-up visit after 1 week of the intervention. Both study visits included collection of anthropometric measures, a fasting blood sample, measures of arterial stiffness, flow-mediated dilation, and endothelial cells via an intravenous catheter.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Euthyroid
* Not currently planning to become pregnant
* Not currently breastfeeding
* No recent history of amenorrhea in the previous 6 months
* Consent to data and specimen banking
* No use of hormonal contraceptives

Inclusion Criteria, type 1 diabetes only:

* Diagnosis of type 1 diabetes for at least 5 years
* On insulin within a year of diagnosis
* Current insulin therapy
* Hemoglobin A1c < 9.5%
* No macroalbuminuria (AER < 200 ug/min)

Inclusion Criteria, non-diabetic controls only:

* Hemoglobin A1c < 5.7%

Exclusion Criteria:

* Pregnant and/or breastfeeding
* Have not had a menstrual cycle in the last 6 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11-24 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation (FMD) at baseline | 1 week
  FMD will be measured following an intravenous saline infusion and ascorbic acid infusion.
Flow-mediated dilation (FMD) at follow-up | 1 week
  FMD will be measured following an intravenous saline infusion and ascorbic acid infusion.
Change in flow-mediated dilation (FMD) | Baseline and 1 week
  FMD will be measured following an intravenous saline infusion and ascorbic acid infusion at baseline and follow-up.
Quantitative immunuofluorescence of endothelial cell proteins at baseline | Baseline
  Expression of estrogen receptor alpha, estrogen receptor beta, endothelial nitric oxide synthase, and phosphorylated endothelial nitric oxide synthase in endothelial cells
Quantitative immunuofluorescence of endothelial cell proteins at follow-up | 1 week
  Expression of estrogen receptor alpha, estrogen receptor beta, endothelial nitric oxide synthase, and phosphorylated endothelial nitric oxide synthase in endothelial cells
Change in quantitative immunuofluorescence of endothelial cell proteins | Baseline and 1 week
  Expression of estrogen receptor alpha, estrogen receptor beta, endothelial nitric oxide synthase, and phosphorylated endothelial nitric oxide synthase in endothelial cells

CONTACTS AND LOCATIONS:
Overall Officials: Janet K Snell-Bergeon, PhD, MPH, Principal Investigator — University of Colorado, Denver